CLINICAL TRIAL: NCT00307307
Title: Magnetic Resonance Characterization of Carotid Atherosclerotic Plaque in Vivo: Effect of High Density Lipoprotein Elevation on Plaque Morphology
Brief Title: Carotid Atherosclerosis Regression at Magnetic Resonance Assessment.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: The Dana Foundation (Other); Merck Sharp & Dohme LLC (Industry); Kos Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CARMA
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Last update posted 2006-05-22 (Estimated); Status verified 2006-03

CONDITIONS: Established Carotid Atherosclerosis
Keywords: atherosclerosis; HDL cholesterol; niacin; MR imaging
MeSH Terms: conditions — Atherosclerosis | interventions — Niacin

INTERVENTIONS:
Drug: Niacin/simvastatin compared to simvastatin alone at 2 doses

SUMMARY:
The primary objective of this randomized, double blind, placebo controlled pilot study is to determine if therapies aimed at lowering LDL cholesterol (HMGCoA reductase inhibitor - simvastatin) or increasing HDL cholesterol (Niaspan) will induce regression of carotid atherosclerotic plaque in vivo using MRI imaging techniques. MR plaque morphology at baseline will be compared to that after 6 and 12 months of therapy and changes in MR characteristics will be compared to changes in lipoprotein parameters and urinary isoprostanes. The effect of moderate LDL reduction, aggressive LDL reduction and the combination of aggressive LDL reduction and HDL elevation on MRI plaque characteristics will be compared by randomly assigning subjects (n=69) with carotid disease (>30% stenosis by ultrasound criteria) to one of three treatment arms;

1. Simvastatin 20 mg daily and placebo Niaspan (n=23)
2. Simvastatin 80 mg daily and placebo Niaspan (n=23)
3. Simvastatin 20 mg daily and active Niaspan (n=23) Treatment group 2 and 3 will have roughly equivalent LDL lowering because of the synergistic LDL lowering effect of the combination of simvastatin and Niaspan.

DETAILED DESCRIPTION:
FULL PROTOCOL

1.0 SYNOPSIS The primary objective of this randomized, double blind, placebo controlled pilot study is to determine if therapies aimed at lowering LDL cholesterol (HMGCoA reductase inhibitor - simvastatin) or increasing HDL cholesterol (Niaspan) will induce regression of carotid atherosclerotic plaque in vivo using MRI imaging techniques. MR plaque morphology at baseline will be compared to that after 6 and 12 months of therapy and changes in MR characteristics will be compared to changes in lipoprotein parameters and urinary isoprostanes. The effect of moderate LDL reduction, aggressive LDL reduction and the combination of aggressive LDL reduction and HDL elevation on MRI plaque characteristics will be compared by randomly assigning subjects (n=69) with carotid disease (>30% stenosis by ultrasound criteria) to one of three treatment arms;

1. Simvastatin 20 mg daily and placebo Niaspan (n=23)
2. Simvastatin 80 mg daily and placebo Niaspan (n=23)
3. Simvastatin 20 mg daily and active Niaspan (n=23) Treatment group 2 and 3 will have roughly equivalent LDL lowering because of the synergistic LDL lowering effect of the combination of simvastatin and Niaspan.

2.0 BACKGROUND Atherosclerotic carotid disease is the largest single etiological factor known to produce focal cerebral ischemia (1). Only a small percentage of patients with asymptomatic carotid atherosclerosis develop stroke but the majority of these have have no warning symptoms. The degree of internal carotid stenosis at ultrasound angiography, the commonest methods of assessing the risk of stroke, are poor predictors of stroke in patients with asymptomatic carotid atherosclerosis (2) and clinical risk factors have a high prevalence but a low relative risk of stroke in these patients. Most plaque rupture occurs in unstable lipid rich plaques with thin fibrous caps weakened by inflammation and apoptosis (3). Thus, the morphological characteristics of carotid plaques may provide important information regarding ischemic risk of carotid lesions. We, and others, are using high resolution MR imaging (4-6) to differentiate carotid plaque elements such as the lipid core, the fibrous cap and hemorrhage with the ultimate goal of determining the ischemic potential of carotid atherosclerotic plaques.

Lipid lowering therapy with statins is considered standard treatment for patients with atherosclerosis and hypercholesterolemia (7-9). Statin therapy reduces LDL cholesterol levels, cardiovascular events and death and retards the progression of atherosclerosis as assessed by noninvasive intima-media thickness (IMT) on carotid ultrasound (10). However, the optimal degree of LDL cholesterol lowering with statins in patients with atherosclerosis remains unclear (7,8) - thus there are a number of ongoing large clinical trials comparing the effect of low dose to high doses of statins on cardiovascular effects in patients with coronary atherosclerosis (eg "Treatment to New Targets"). Low HDL cholesterol is an independent risk factor for the development and progression of atherosclerosis (11). Niacin is one of a few effective therapies that significantly elevates HDL levels and was shown to reduce cardiovascular events in patients with known coronary atherosclerosis prior to the development of statin drugs (12,13). Increased HDL is thought to promote reverse cholesterol transport from the peripheral tissues including atherosclerotic plaque (14-16). Presently, niacin is not considered standard therapy in patients with known atherosclerosis. Niaspan is a new controlled-release form of niacin that is administered once daily, is better tolerated than crystalline niacin which is given 3 times a day (17,18). It has been shown to result in a greater than 30% increase in HDL cholesterol and preliminary data suggest that it is safe and effective and not associated with hepatotoxicity (19). In the proposed study patients (n=60) with carotid disease (>30% stenosis by ultrasound criteria) will be randomly assigned to one of three treatment arms;

1. Simvastatin 20 mg daily and placebo Niaspan (n=23)
2. Simvastatin 80 mg daily and placebo Niaspan (n=23)
3. Simvastatin 20 mg daily and active Niaspan (n=23) Thus, the effect of Simvastatin 10 mg (moderate LDL reduction), Simvastatin 80 mg (aggressive LDL reduction) and the combination of Simvastatin and Niaspan (aggressive LDL reduction and HDL elevation) on MRI plaque characteristics will be compared.

3.0 OBJECTIVES

The primary objective of this randomized, double blind, placebo controlled pilot study is to determine if therapies aimed at lowering LDL cholesterol (HMGCoA reductase inhibitors - statins) or increasing HDL cholesterol (Niaspan) will induce regression of carotid atherosclerotic plaque in vivo using MRI imaging techniques. MR plaque morphology at baseline will be compared to that after 6 and 12 months of therapy and changes in MR characteristics will be compared to changes in lipoprotein parameters and urinary isoprostanes.

3.1 Primary End-Point The primary end-point is the change in carotid plaque volume at MRI after 12 months of treatment.

3.2 Secondary End-Points

1. - change in carotid plaque lipid content at MRI after 12 months
2. - change in lipid parameters after 12 months
3. - change in urinary isoprostane excretion after 12 months

4.0 STUDY DESIGN

4.1 Description

This study will be randomized, double-blind and placebo controlled. Sixty patients will be randomly assigned to (1) Simvastatin 20 mg and placebo Niaspan, (2) Simvastatin 80 mg and placebo Niaspan or (3) Simvastatin 20 mg and active Niaspan. The study will involve 6 outpatient visits to the General Clinical Research Center (GCRC) at the Hospital of the University of Pennsylvania. Each visit will last approximately 2 hours.

4.2 Number of Subjects

Sixty nine (69) subjects with known carotid atherosclerosis will be investigated.

5.0 STUDY POPULATION

Source of subjects

Subjects with carotid disease, identified on (1) routine carotid ultrasound examinations at the vascular laboratories of the University of Pennsylvania Health System and VA Medical Center, and (2) through local advertisement will be invited to participate in the study. Subjects will be contacted by letter inviting them to participate in the study. Subjects will be screened according to the following inclusion and exclusion criteria;

Inclusion Criteria Age >18 and <90 years Capacity for giving written informed consent Carotid stenosis of >30% by ultrasound criteria LDL cholesterol level of >100mg/dl Systolic BP < 170 and diastolic BP < 100 under resting conditions Negative pregnancy test if female of child-bearing potential

Exclusion criteria Recent (< 3 months) history of stroke, transient ischemic attack, myocardial infarction, unstable angina or critical limb ischemia, Contraindications to MRI (claustrophobia, presence of pacemakers, defibrillators, metal foreign bodies), History of side effect/adverse reaction on HMGCoA reductase inhibitor, Niaspan or niacin, Poorly controlled diabetes (HbA1c >8%), History of myositis, liver disease or abnormal LFTs, Need for combination therapy for the control of severe hyperlipidemia, Abnormal LFT (>2 fold upper limit normal), Active infection or malignancy.

6.0 STUDY PROCEDURES The study will involve 6 outpatient visits to the General Clinical Research Center (GCRC) at the Hospital of the University of Pennsylvania. Each visit will last approximately 2 hours.

6.1 Pre-treatment Period All subjects will be asked to come to GCRC for a screening visit. During this visit, a complete medical history and physical examination will be performed. Dosage of all chronic medication will be recorded. Supine resting blood pressure, an electrocardiogram and the following fasting routine laboratory studies will be performed; Hematology; hemoglobin, hematocrit, MCV, white blood count and platelet count Blood chemistries; sodium, potassium, chloride, creatinine, fasting glucose, albumin, alkaline phosphatase, total bilirubin, AST, ALT, uric acid total cholesterol, LDL, HDL, triglycerides lipoprotein (a) and HbA1c.

Urinalysis Urinary HCG - for women of child bearing potential. Eligible subjects will undergo a full dietary assessment by the GCRC research dietician using a quantitative questionnaire. Subjects will be instructed to comply with recommended AHA dietary guidelines so that dietary intake of macronutrients including fat and cholesterol will be similar across all subjects. Dietary compliance will be monitored at baseline and each study visit by 24-hour recall of dietary intake. The Dietary Analysis System (DIETSYS) will be used to analyze the food frequency questionnaires and the Food Processor Plus (ver 6.0) will be used to analyze dietary recalls.

6.2 Concurrent Treatment The use of most concurrent medications will not be restricted during the study period. Indeed, aspirin use and antihypertensive therapies will be encouraged when appropriate. Lipid lowering medications, other than those in the study will be stopped prior to randomization. For example all HMGCoA reductase inhibitors will be replaced by simvastatin at the time of randomization.

6.3 Treatment Period Eligible subjects will be asked to collect a 12-hour urine sample prior to randomization and bring them to the GCRC on the morning of randomization where they will be processed and stored until analysis. Baseline blood samples will be collected for hematology, chemistry and lipoprotein analysis as per screening. Subjects will undergo micro MRI scans of the carotid arteries in the MRI center adjacent to the GCRC. A subset of volunteers (n=10) will be asked to undergo a second baseline MRI scan within a week of the first scan in order to determine the reproducibility of the quantitative MRI technique. Subjects will then be randomized in a double blind manner to (1) Simvastatin 20 mg and placebo Niaspan, (2) Simvastatin 80 mg and placebo Niaspan or (3) Simvastatin 20 mg and active Niaspan. Simvastatin tablets will be provided by Merck Pharmaceuticals, the manufacturer of Simvastatin. Niaspan tablets (500mg) and matching placebo will be provided by KOS, the company that manufactures Niaspan. Niaspan will be titrated according to clinical guidelines - 500 mg at bedtime for 1 month, 1000 mg at bedtime for the next month and finally 2000 mg at bedtime for the rest of the study. At the randomization visit, these specific instructions for titration of Niaspan or placebo (given in matching tablets in an identical way) will be discussed and given to each subject with a one-month supply of study drug.

Both Niaspan (KOS Pharmaceuticals) and simvastatin (Zocor; Merck Pharmaceuticals) are commercially available drugs that are FDA approved for management of hyperlipidemia at the doses, formulation and route of administration proposed in this study.

Return visits will be scheduled for 1, 3, 6 and 12 months. At each of these visits history, physical exam and blood testing (hematology, chemistry, fasting lipoproteins) will be undertaken. In addition, urine collections and MRI studies will be performed at 6 and 12 months. Known adverse effects, such as flushing and muscle cramps will be screened for at each visit. Subjects will be discontinued from the study for the following reasons;

1. intolerable side effects from the study medications
2. increase in either ALT or AST greater than 3 times upper limit of normal
3. HbA1c>9%
4. uric acid >11.0
5. pregnancy

Eligible subjects will be asked to increase study medication to 2000mg daily at bedtime after the second month. Every attempt will be made to titrate the Niaspan/placebo to 2000mg per day, but if this is not possible the subject will be maintained on the maximal achievable dose. The duration of the study is 12 months. All assessments will be made by personnel blinded to the study treatment.

6.4 Duration of the Study The duration of the entire study will be approximately 18 months. Actual study drug treatment will be of 12 months duration. Each subject will undergo screening approximately 2 weeks prior to randomization and it is anticipated that subjects will be enrolled over a 6 month period.

6.5 Premature Withdrawal from the Study

A volunteer may be withdrawn from the trial for the following reasons:

* Any adverse event thought to warrant withdrawal by the investigator,
* Poor compliance thought to warrant withdrawal by the investigator,
* Volunteer's desire to withdraw from the study at any time,
* Protocol or entry criteria violation,
* Pregnancy.

The reasons for withdrawal and the final outcome in cases of adverse events will be documented on the Case Report Form. Subjects who do not complete the study will be replaced.

7.0 EFFICACY ASSESSMENT

7.0 Variables to be measured for Efficacy Assessment Magnetic Resonance Imaging of Carotid Atherosclerotic Plaques: A variety of MRI techniques have been optimized to permit sufficient resolution to determine size and composition of atherosclerotic plaque. These include "black-blood" imaging techniques, fast spin echo sequences, and fat suppression techniques in addition to customized coils (4-6). Customized surface coils will be constructed to further improve the signal-to-noise ratio. While the coils and some of the sequences are not FDA approved as they are custom built, they all fall under the category of "non-significant risk devices". These techniques have already been established for this purpose at the MRI center at the Hospital of the University of Pennsylvania. The imaging protocol consists of a combination of black blood (fast spin echo and double inversion recovery fast spin echo sequences) and bright blood imaging (time-of-flight MRA sequence) to achieve optimal contrast between the arterial lumen and the vessel wall. Specifically, the following sequences are obtained: (1) 3D time of flight (TOF) MRA of the carotid bifurcation; (2) axial T1-weighted fast spin echo; (3) axial proton density-weighted weighted double inversion recovery fast spin echo (DIR-FSE) through plaque; and (4) axial T2-weighted weighted DIR-FSE through plaque. Total plaque volume will be quantified as follows;

Plaque volume = (computer assisted calculation of region of interest-ROI) x (slice thickness) x (no. of slices).

Plaque composition will be estimated using established imaging criteria for the 4 image contrast weightings (Table 1).

Table 1 Criteria used for identification of plaque constituents. TOF T1-W PD-W T2-W Calcification Low Low Low Low Hemorrhage High High/Moderate Variable Variable Lipid core Moderate High High Variable Fibrous cap Moderate/Low Moderate High Variable Note: Intensity descriptors are relative to intensity of sternocleidomastoid muscle.

Lipoprotein Determination: Total cholesterol, LDL cholesterol, HDL cholesterol, lipoprotein (a) and triglyceride levels will be determined by standardized techniques in the routine chemistry laboratory of the Hospital of the University of Pennsylvania.

Urinary Isoprostanes: Urinary isoprostanes will be measured by mass spectrometry / gas chromatography (GC / MS) as previously described by the PI (20). Following the addition of a deuterated isoprostane internal standard, urine samples are extracted from the aqueous matrix by solid phase extraction techniques, purified by thin layer chromatography, derivatized, and analyzed by GC / MS in the negative ion chemical ionization (NICI) mode. Quantification is accomplished by taking the ratio of the area under the peak of the ion representing the endogenous compound to that of the internal standard.All subjects who complete the study will be considered evaluable for efficacy assessment.

7.2 Criteria for Evaluability of Efficacy Assessment

All subjects who complete the study will be considered evaluable for efficacy assessment.

8.0 SAFETY ASSESSMENT

8.1 Variables to be Measured for Safety Assessment

Safety measures to be monitored include

1. symptoms (flushing, abdominal pain, tiredness)
2. transaminases
3. HbA1c
4. uric acid

8.2 Criteria for Evaluability of Safety Assessment

All subjects entered into the trial will be considered evaluable for safety assessment.

9.0 STATISTICAL CONSIDERATIONS

There is currently no data available on the effect of therapies on carotid atherosclerotic plaque morphology using MRI on which to base sample size estimations. Therefore, sample sizes are based on the desire to acquire pilot data to allow the determination of the actual numbers required for a study examining both MR characteristics and clinical endpoints. A sample size of 69 (23 subjects per arm) will provide 80% power to detect the hypothesized difference (15%) in the primary endpoint (plaque volume) between 2 different treatment arms at an alpha of 0.05. The number of subjects needed for future full-scale clinical studies will be dependent on the coefficient of variation of repeated baseline quantitative MRI scans and the change in plaque volume (primary end-point) following an intervention. These parameters will be defined by the proposed pilot study.

10.0 DATA COLLECTION, MONITORING AND AE REPORTING

10.1 Case Report Forms

Case Report Forms (CRFs) will be provided for each subject. Subjects must not be identified by name on any study documents. Subjects will be identified by the Patient Identification Number (PIN) and Study Identification Number (SID). All data on the CRF will be legibly recorded in black ink or typed. Corrections will be made by striking the incorrect entry with a single line through it and then adding the correct information adjacent to it. The corrections will be initialed and dated by the investigator or designated qualified individual. Any requested information that is not obtained as specified in the protocol will be indicated on the CRFs as "not done" (ND) or "not applicable" (NA).

10.2 Data Management

The CRF design and data management will be performed by the PI and research assistants.

10.3 Monitoring

The PI will review the research records for accuracy, completeness and legibility. The investigator or designated qualified individual will make study documents (eg consent forms, drug distribution forms, case report forms) and pertinent hospital or clinic records available for inspection by the Food and Drug Administration (FDA) for conformation of the data.

10.4 Adverse Experience (AE) Reporting

Adverse Experiences (AEs) will be monitored throughout the study and such events will be recorded on the Adverse Experience Case Report Forms. An AE is defined as any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with the use of the study medication, whether or not considered related to the use of the product. The AEs will be graded on a three-point scale (mild, moderate severe) and a drug relationship assigned.

Any serious or unexpected adverse events will be reported within 24 hours to the FDA and the IRB of the University of Pennsylvania. Adverse events are defined as serious when they are fatal, life-threatening or result in in-patient hospitalization or prolongation of hospitalization. In addition the occurrence of malignancy is always considered serious adverse advents. Adverse events are considered unexpected if their occurrence, or severity or frequency have not been previously reported in concomitance with Niaspan or HMGCoA reductase inhibitor therapy.

11.0 ETHICAL CONSIDERATIONS

11.1 Institutional Review Board (IRB)

The study protocol will be reviewed by the committee on Studies involving Human Beings at the University of Pennsylvania. A copy of the letter of approval and correspondence with the IRB will be retained by the investigators.

11.2 Informed Consent

Written informed consent will be obtained from every volunteer participating in the study after adequate explanation of the object of the study and possibly adverse effects of the drug treatment.

11.3 Subject Confidentiality

The medical information gathered during this study will be treated confidentially except as may be required by law. Regulatory authorities, including the US Food and Drug Administration, might review the medical records to verify the accuracy of the information collected. Subjects will not be identified by name on any study documents and, if the results are published the subjects' identity will not be disclosed.

REFERENCES

1. Gelabert HA and Moore WS. Carotid endarterectomy: current status. Curr Prob Surg 1991; XXVIII: 187-262.
2. Moneta GL, Taylor DC, Zierler RE, Kazmers A, Beach K and Stradness DE. Asymptomatic high grade internal carotid carotid artery stenosis: is stratification according to risk factors or duples spectral analysis possible. J Vasc Surg 1989; 10: 475.
3. Libby P, Li H. Vascular cell adhesion molecule-1 and smooth muscle cell activation during atherogenesis. J Clin Invest 1993; 92: 538-539
4. Skinner MP, Yuan C, Mitsumori L, Hayes CE, Raines EW, Nelson JA, Ross R. Serial magnetic-resonance imaging of experimental atherosclerosis detects lesion fine structure, progression and complications in vivo. Nature Medicine 1995; 1: 69-73.
5. Toussaint J-F, Southern JF, Fuster V, Kantor HL. T2-weighted contrast for NMR characterization of human atherosclerosis. Arterioscler Thromb Vasc Biol 1995; 15: 1533-42.
6. Toussaint J-F, LaMuraglia GM, Southern JF, Fuster V, Kantor HL. Magnetic resonance images lipid, fibrous, calcified hemorrhagic and thrombotic components of human atherosclerosis in vivo. Circulation 1996; 94: 932-938.
7. Scandinavian Simvastatin Survival Study Group. Randomized trial of cholesterol lowering in 4444 patients with coronary heart disease: the Scandinavian Simvastatin Survival Study (4S). Lancet 1994; 344: 1383-89.
8. Ridker, P. M., N. Rifai, M. A. Pfeffer, F. M. Sacks, L. A. Moye, S. Goldman, G. C. Flaker, and E. Braunwald. Inflammation, pravastatin, and the risk of coronary events after myocardial infraction in patients with average cholesterol levels. Cholesterol and recurrents events (CARE) investigatiors . Circulation 1998; 98:839-844.
9. Jukema JW, Bruschke AVG, van Boven AJ et al; on behalf of the REGRESS Study Group. Effects of lipid lowering by pravastatin on progression and regression of coronary artery disease in symptomatic men with normal to moderately elevated serum cholesterol levels. The regression growth evaluation statin study (REGRESS). Circulation 1995; 91: 2528-40.
10. Crouse JR, Byington RP, Bond MG, Espeland MA, Craven TE, Sprinkle JW, McGovern ME, Furberg CD. Pravastatin, lipids and atherosclerosis in the carotid arteries (PLAC-II). Am J Cardiol 1995;75: 455-9.
11. Vega, G. L. and S. M. Grundy. Hypoalphalipoproteinemia (low high density lipoprotein) as a risk factor for coronary heart disease. Curr. Opin. Lipidol. 1996; 7:209-216.
12. Canner, P. L., K. G. Berge, N. K. Wenger, J. Stamler, L. Friedman, R. J. Prineas, and W. Friedwald. Fifteen year mortality in Coronary Drug Project patients: Long term benefit with niacin. J Am Coll Cardiol 1986; 8:1245-1255.
13. Blankenhorn DH, Nessim SA, Johnson RL, Sanmarco ME, Azen SP, Cashin-Hemphill L. Beneficial effects of colestipol-niacin therapy on coronary atherosclerosis and coronary venous bypass grafts. JAMA 1987; 257: 3233-3240.
14. Reichl, D. and N. E. Miller. Pathophysiology of reverse cholesterol transport. Insights from inherited disorders of lipoprotein metabolism. Arteriosclerosis 1989; 9: 785-797.
15. Plump AS, Scott CJ, Breslow JL. Human apolipoprotein A-I gene expression increases high density lipoprotein and suppresses atherosclerosis in the apolipoprotein E-deficient mouse. Proc Natl Acad Science 1994; 91: 9607-9611.
16. Eriksson M, Carlson LA, Miettinen TA, Angelin B. Stimulation of fecal steroid excretion after infusion of recombinant proapolipoprotein A-I. Potential reverse cholesterol transport in humans. Circulation 1999; 100: 594-598.
17. Rosenson, R. S. 1993. Low levels of high-density lipoprotein cholesterol (hypoalphalipoproteinemia): an approach to management. Arch Intern Med 1993; 153:1528-1538.
18. Alderman JD, Pasternak RC, Sacks FM, Smith HS, Monrad ES, Grossman W. Effect of a modified, well tolerated niacin regimen on serum total cholesterol, high density lipoprotein and the cholesterol to high density lipoprotein ratio. Am J Cardiol 1989; 64: 725-729.
19. Morgan, J. M., D. M. Capuzzi, J. R. Guyton, R. M. Centor, R. Goldberg, D. C. Robbins, D. Dipette, S. Jenkins, and S. Marcovina. Treatment effect of Niaspan, a controlled-release niacin, in patients with hypercholesterolemia: a placebo-controlled trial. J Cardiovasc Pharm Ther 1996; 1:195-202.
20. Reilly MP, Pratico D, Delanty N, DiMinno G, Tremoli E, Rader D, Kapoor S, Lawson JA, Rokach J, FitzGerald GA. Increased biosynthesis of distinct F2-isoprostanes in hypercholesterolemia. Circulation 1998; 98: 2822-2828.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 90 years
* Capacity for giving written informed consent
* Carotid stenosis of > 30% by ultrasound criteria
* LDL cholesterol level of > 100mg/dl
* Systolic BP < 170 and diastolic BP < 100 under resting conditions
* Negative pregnancy test if female of child-bearing potential

Exclusion Criteria:

* Recent (< 3 months) history of stroke, transient ischemic attack, myocardial infarction, unstable angina or critical limb ischemia
* Contraindications to MRI (claustrophobia, presence of pacemakers, defibrillators, metal foreign bodies)
* History of side effect/adverse reaction on HMGCoA reductase inhibitor
* Niaspan or niacin
* Poorly controlled diabetes (HbA1c > 8%)
* History of myositis, liver disease or abnormal LFTs
* Need for combination therapy for the control of severe hyperlipidemia
* Abnormal LFT (> 2 fold upper limit normal)
* Active infection or malignancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69
Dates: Start 2000-01; Study Completion 2005-09

PRIMARY OUTCOMES:
Change in MRI estimates of carotid atherosclerosis

SECONDARY OUTCOMES:
Change in lipoproteins and inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Muredach P Reilly, MB MSCE, Principal Investigator — University of Pennsylvania